CLINICAL TRIAL: NCT02511067
Title: Evaluation Of the Safety, Tolerability and Efficacy of Ranibizumab and Tocilizumab in Eyes With Diabetic Macular Edema.
Brief Title: Ranibizumab for Edema of the mAcula in Diabetes: Protocol 4 With Tocilizumab: The READ-4 Study
Acronym: READ-4
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding lost and study never started
Sponsor: University of Nebraska (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 0594-15-FB
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — tocilizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ranibizumab 0.3 mg (Active Comparator): Mandatory monthly treatments with Intravitreal (IVT) ranibizumab (0.3 mg) starting at Baseline (BL) until Month 6. Starting at Month 6, treatments will be administered on as-needed basis, based on retreatment criteria.
  Interventions: Drug: Ranibizumab
- Tocilizumab (8.0 mg/kg) (Experimental): Mandatory monthly Intravenous (IV) infusions with tocilizumab (8.0 mg/kg) starting at Baseline (BL) until Month 6. Starting at Month 6, treatments will be administered on as-needed basis with IVT ranibizumab (0.3 mg), based on the retreatment criteria.
  Interventions: Drug: Tocilizumab
- Tocilizumab (8.0 mg /kg) plus Ranibizumab 0.3 mg (Experimental): Mandatory Intravitreal (IVT) ranibizumab 0.3 mg at Baseline (BL) followed with an IV infusion of tocilizumab (8.0 mg/kg) on same day starting at Baseline (BL) until Month 6. Combination treatments (IVT ranibizumab 0.3 mg followed by IV tocilizumab 8.0 mg/kg infusion administered at same visit) will be given every month until Month 6. Starting at Month 6, treatments will continue to be administered on as-needed basis with IVT ranibizumab (0.3 mg), based on retreatment criteria.
  Interventions: Drug: Tocilizumab; Drug: Ranibizumab

INTERVENTIONS:
Drug: Tocilizumab — Intravenous Infusion of Tocilizumab ( 8.0 mg/kg)
  Other Names: Actemra
  Arms: Tocilizumab (8.0 mg /kg) plus Ranibizumab 0.3 mg; Tocilizumab (8.0 mg/kg)
Drug: Ranibizumab — Intravitreal injection of Ranibizumab (0.3mg)
  Other Names: Lucentis, Susvimo
  Arms: Ranibizumab 0.3 mg; Tocilizumab (8.0 mg /kg) plus Ranibizumab 0.3 mg

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and efficacy of Ranibizumab and Tocilizumab alone and in combination in eyes with Diabetic Macular Edema.

DETAILED DESCRIPTION:
This study will evaluate the safety of intravenous (IV) infusions of Tocilizumab in the treatment of subjects with diabetic macular edema (DME) as monotherapy and in combination with intravitreal (IVT) Ranibizumab. It will also evaluate the percentage change in central retinal thickness (CRT) from baseline (BL) to Month 6 in the study eye as assessed by spectral-domain optical coherence tomography (SD-OCT). Other study objectives are to determine: the change in visual acuity (VA) from baseline to Months 3, 6 and 12, the change in CRT from baseline to Months 3, 6 and 12 in all the three treatment arms and determine the number of eyes requiring rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent and authorization of use and disclosure of protected health information

  * Age ≥18 years
  * Diagnosis of diabetes mellitus (type 1 or type 2)
  * Serum HbA1c ≥ 5.5% and ≤10% within 12 months of randomization. (It is important to be certain that the patients in the READ-4 Study have diabetes, which will suggest that the macular edema is secondary to diabetes. The American Diabetes Association has suggested that a HbA1c ≥ 5.5% may suggest the presence of diabetes mellitus.)
  * Have diabetic macular edema (DME) with central subfield thickness of ≥ 310 microns on spectral domain optical coherence tomography (SD-OCT).
  * Retinal thickening secondary to diabetes mellitus involving the center of the fovea (centered-involved macular edema).
  * Best corrected visual acuity score in the study eye of 20/32 to 20/400 inclusive (Snellen equivalents using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at a distance of 4 meters). If both eyes are eligible, the investigator will select the eye to be enrolled as the study eye. There is no specific visual acuity requirement for the fellow eye at time of study eye enrollment. However, if the fellow eye is to receive ranibizumab, it must have an entry visual acuity of 20/32 to 20/400 inclusive (Snellen equivalents using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at a distance of 4 meters) at the time of the initial treatment.
  * In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from diabetic macular edema (DME) and not from other obvious causes of decreased vision.
  * Female of childbearing potential must have a negative serum pregnancy test within 28 days of randomization
  * Females of child-bearing potential may participate in this trial only if using a reliable means of contraception (e.g. physical barrier (patient and partner), contraceptive pill or patch, spermicide and barrier, or intrauterine device (IUD))
  * If a non-sterile male, commitment to the use of effective contraception (birth control) for the duration of the study is necessary.

Exclusion Criteria:

* • Panretinal photocoagulation or macular photocoagulation within 90 days prior to Day 0 in the study eye.

  * Presence of active proliferative diabetic retinopathy
  * Use of any intravitreal injections (including but not limited to anti vascular endothelial growth factor therapy or steroids) within 60 days prior to Day 0 in the study eye.
  * Use of Tocilizumab (IV or SC) within 180 days prior to Day 0.
  * Use of intravitreal dexamethasone implant within 120 days (4 months) prior to Day 0 in the study eye.
  * Use of intravitreal triamcinolone within 120 days prior to Day 0 in the study eye.
  * Use of intravitreal fluocinolone implant within 3 years (36 months) prior to Day 0 in the study eye.
  * Intraocular surgery within 90 days prior to Day 0 in the study eye
  * History of vitrectomy in study eye
  * Capsulotomy within 30 days prior to Day 0 in the study eye
  * Any planned ocular surgery (including cataract extraction or capsulotomy) of the study eye anticipated within the first 180 days following Day 0;
  * Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye;
  * Media opacity that would limit clinical visualization;
  * Presence of any form of ocular malignancy in the study eye, including choroidal melanoma
  * History of herpetic infection in the study eye or adnexa
  * Presence of known active or inactive toxoplasmosis in either eye
  * Ocular or periocular infection in either eye
  * Participation in other investigational drug or device clinical trials within 30 days prior to Day 0, or planning to participate in other investigational drug or device clinical trials within 180 days following Day 0. This includes both ocular and non-ocular clinical trials.
  * Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
  * Prior treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20.
  * Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
  * Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
  * Any previous treatment with tocilizumab.
  * Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.

Concurrent Ocular Conditions

* Proliferative diabetic retinopathy in the study eye, with the exceptions of

  . Inactive, fibrotic proliferative diabetic retinopathy that has regressed following panretinal laser photocoagulation
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by optical coherence tomography (OCT).
* Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), macular ischemia, or organized hard exudate plaque
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., Age-related macular degeneration (AMD), ocular histoplasmosis, or pathologic myopia).
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the first 6-month study period
* Cataract surgery in the study eye within 3 months of study entry; Yttrium-Aluminum-Garnet (YAG) laser capsulotomy within 1 month of study entry; or any other intraocular surgery within 3 months preceding Day 0.
* History of vitreoretinal surgery in the study eye within 3 months of study entry
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 30 mm) Hg despite treatment with anti-glaucoma medications)

Systemic Conditions or Exclusions for General Safety:

* Uncontrolled diabetes mellitus, as evidenced by glycosylated hemoglobin (HbA1c) value >10%
* Blood pressure exceeding 180/100 (sitting) during the screening period
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
* Have a history of hypersensitivity to ranibizumab or any of their components
* Presence of any ulcerative wounds
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal (including dialysis), hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease
* History of diverticulitis, diverticulosis requiring antibiotic treatment or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis or other symptomatic lower GI conditions that might predispose to perforations.
* Current active liver disease as determined by principal investigator
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Active Tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be screened for latent Tuberculosis (TB) and, if positive, treated following local practice guidelines prior to initiating tocilizumab. Patients treated for tuberculosis with no recurrence in 3 years are permitted.
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured)
* Pregnant women or nursing (breast feeding) mothers.
* Patients with reproductive potential not willing to use an effective method of contraception.
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Patients with lack of peripheral venous access.

Laboratory Exclusion Criteria:

Subjects who meet any of the following laboratory criteria at screening should not be enrolled in the study unless the values have normalized. In addition, if any study subject meets any of the following criteria during the course of the study, the investigator can consider withholding treatment (tocilizumab and/or ranibizumab) at particular visits and initiating appropriate management, and can resume treatment with study drugs at subsequent visits once the laboratory values have normalized or once the investigator have considered that it is safe to resume therapy.

* INR ≥ 3.0 (e.g. due to current treatment with warfarin). The use of aspirin or other anticoagulants is not an exclusion
* Serum creatinine > 1.4 mg/dL (124 μmol/L) in female patients and > 1.6 mg/dL (141 μmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total Bilirubin > ULN
* Platelet count < 100 x 109/L (100,000/mm3)
* Hemoglobin < 8.5 g/L (8.5 g/dl; 5.3 mmol/L)
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* Positive Hepatitis HBsAg, or Hepatitis C antibody

Other:

* Inability to comply with study or follow-up procedures
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  To evaluate the safety of IV infusions of tocilizumab in treatment of subjects with diabetic macular edema (DME) as monotherapy and in combination with Ranibizumab
Anatomic Retinal Changes | Month 6
  To evaluate the percentage change in central retinal thickness (CRT) from Baseline to Month 6 in the study eye as assessed by spectral domain-optical coherence tomography (SD-OCT).

SECONDARY OUTCOMES:
Visual Acuity | Month 3, 6, and 12
  Change in visual acuity (VA) from baseline to months 3, 6 and 12
Anatomic Retinal Changes | Month 3, 6, and 12
  Percentage change in change in central retinal thickness (CRT) from baseline to months 3, 6 and 12 in all the three treatment arms
Rescue Therapy | Month 6
  Number of eyes requiring rescue therapy

CONTACTS AND LOCATIONS:
Overall Officials: Diana Do, MD, Principal Investigator — University of Nebraska

REFERENCES:
- [Background] Bourne RR, Stevens GA, White RA, Smith JL, Flaxman SR, Price H, Jonas JB, Keeffe J, Leasher J, Naidoo K, Pesudovs K, Resnikoff S, Taylor HR; Vision Loss Expert Group. Causes of vision loss worldwide, 1990-2010: a systematic analysis. Lancet Glob Health. 2013 Dec;1(6):e339-49. doi: 10.1016/S2214-109X(13)70113-X. Epub 2013 Nov 11. PMID 25104599
- [Background] Klein R. Hyperglycemia and microvascular and macrovascular disease in diabetes. Diabetes Care. 1995 Feb;18(2):258-68. doi: 10.2337/diacare.18.2.258. PMID 7729308
- [Background] Nguyen QD, Tatlipinar S, Shah SM, Haller JA, Quinlan E, Sung J, Zimmer-Galler I, Do DV, Campochiaro PA. Vascular endothelial growth factor is a critical stimulus for diabetic macular edema. Am J Ophthalmol. 2006 Dec;142(6):961-9. doi: 10.1016/j.ajo.2006.06.068. Epub 2006 Aug 2. PMID 17046701
- [Background] Koskela UE, Kuusisto SM, Nissinen AE, Savolainen MJ, Liinamaa MJ. High vitreous concentration of IL-6 and IL-8, but not of adhesion molecules in relation to plasma concentrations in proliferative diabetic retinopathy. Ophthalmic Res. 2013;49(2):108-14. doi: 10.1159/000342977. Epub 2012 Dec 18. PMID 23257933
- [Background] Sonoda S, Sakamoto T, Yamashita T, Shirasawa M, Otsuka H, Sonoda Y. Retinal morphologic changes and concentrations of cytokines in eyes with diabetic macular edema. Retina. 2014 Apr;34(4):741-8. doi: 10.1097/IAE.0b013e3182a48917. PMID 23975003
- [Background] Treatment techniques and clinical guidelines for photocoagulation of diabetic macular edema. Early Treatment Diabetic Retinopathy Study Report Number 2. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1987 Jul;94(7):761-74. doi: 10.1016/s0161-6420(87)33527-4. PMID 3658348
- [Background] Boyer DS, Yoon YH, Belfort R Jr, Bandello F, Maturi RK, Augustin AJ, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Three-year, randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with diabetic macular edema. Ophthalmology. 2014 Oct;121(10):1904-14. doi: 10.1016/j.ophtha.2014.04.024. Epub 2014 Jun 4. PMID 24907062
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Arevalo JF. Diabetic macular edema: changing treatment paradigms. Curr Opin Ophthalmol. 2014 Nov;25(6):502-7. doi: 10.1097/ICU.0000000000000102. PMID 25211039
- [Background] Chun DW, Heier JS, Topping TM, Duker JS, Bankert JM. A pilot study of multiple intravitreal injections of ranibizumab in patients with center-involving clinically significant diabetic macular edema. Ophthalmology. 2006 Oct;113(10):1706-12. doi: 10.1016/j.ophtha.2006.04.033. PMID 17011952
- [Background] Do DV, Nguyen QD, Khwaja AA, Channa R, Sepah YJ, Sophie R, Hafiz G, Campochiaro PA; READ-2 Study Group. Ranibizumab for edema of the macula in diabetes study: 3-year outcomes and the need for prolonged frequent treatment. JAMA Ophthalmol. 2013 Feb;131(2):139-45. doi: 10.1001/2013.jamaophthalmol.91. PMID 23544200
- [Background] Mesquida M, Molins B, Llorenc V, Sainz de la Maza M, Adan A. Long-term effects of tocilizumab therapy for refractory uveitis-related macular edema. Ophthalmology. 2014 Dec;121(12):2380-6. doi: 10.1016/j.ophtha.2014.06.050. Epub 2014 Sep 6. PMID 25204610
- [Background] Funatsu H, Yamashita H, Ikeda T, Mimura T, Eguchi S, Hori S. Vitreous levels of interleukin-6 and vascular endothelial growth factor are related to diabetic macular edema. Ophthalmology. 2003 Sep;110(9):1690-6. doi: 10.1016/S0161-6420(03)00568-2. PMID 13129863
- [Background] Shimizu E, Funatsu H, Yamashita H, Yamashita T, Hori S. Plasma level of interleukin-6 is an indicator for predicting diabetic macular edema. Jpn J Ophthalmol. 2002 Jan-Feb;46(1):78-83. doi: 10.1016/s0021-5155(01)00452-x. PMID 11853719
- See also: Study of the Safety, Tolerability, and Bioactivity of Tocilizumab On Patients With Non-infectious UVEITIS: The STOP-UVEITIS Study. NCT01717170. — https://clinicaltrials.gov/